CLINICAL TRIAL: NCT03492203
Title: Remote Cognitive Remediation for Depression
Acronym: RECORD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Christopher Bowie, Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSYC-189-16
Record Dates: First submitted 2016-12-24; First posted 2018-04-10 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Major Depression
Keywords: Cognitive Remediation; Neurocognition; Severe mental illness; Remote treatment
MeSH Terms: conditions — Depressive Disorder, Major; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Cognitive Remediation -Long-term (Experimental): Participants in the long-term treatment will receive 24 weeks of active cognitive remediation. Participants will complete 24 weeks of on-line computer exercises and participate in an on-line forum to facilitate strategy monitoring and bridging strategies.
  Interventions: Behavioral: Active Cognitive Remediation; Behavioral: Online computer exercises; Behavioral: Strategy monitoring; Behavioral: Bridging strategies
- Active Cognitive Remediation -Short-term (Active Comparator): Participants in the short-term treatment will receive 12 weeks of active cognitive remediation (the standard length of time in the literature). Participants will complete 12 weeks of on-line computer exercises and participate in an on-line forum to facilitate strategy monitoring and bridging strategies.
  Interventions: Behavioral: Active Cognitive Remediation; Behavioral: Online computer exercises; Behavioral: Strategy monitoring; Behavioral: Bridging strategies
- Cognitive Remediation Control (Placebo Comparator): Participants in the comparison training group will login to the same training environment but the cognitive load will not adjust as it does in the experimental conditions. Participants in this group will complete 12 weeks of on-line computer exercises.
  Interventions: Behavioral: Cognitive Remediation Control; Behavioral: Online computer exercises; Behavioral: Strategy monitoring; Behavioral: Bridging strategies

INTERVENTIONS:
Behavioral: Active Cognitive Remediation — Cognitive remediation engages participants in computerized exercises meant to improve cognitive functions and provides therapist feedback for how these improvements manifest in everyday life. The novel components of CR in this study will be the delivery of treatment remotely.
  Arms: Active Cognitive Remediation -Long-term; Active Cognitive Remediation -Short-term
Behavioral: Cognitive Remediation Control — The investigators have developed a 'comparison' cognitive remediation treatment in collaboration with the same company that produced the cognitive exercises. These procedures include the same stimuli but are adjusted without increasing cognitive load.
  Arms: Cognitive Remediation Control
Behavioral: Online computer exercises — There are 30 unique cognitive exercises in the program (sbtpro.com). The investigators will prescribe 24 exercises in the domains most commonly impaired in MDD: six targeting executive functions, ten targeting memory, and eight targeting attention and working memory. The specific activities are prescribed in a fixed, systematic order, such that the participants have a schedule of exercises that address several different cognitive domains each week and return to exercises in subsequent weeks. Parameters are automatically adjusted based on participant performance across 30 difficulty levels. Participants are prescribed two 20-minute sessions per day, five days per week, for the duration of the study.
Behavioral: Strategy monitoring — Therapists communicate with participants in asynchronous private and group forums, where specific responses to questions prime flexible strategy formation, monitoring of strategies, and bridging to real world functioning. Participants use logs to track their own strategies and upload this information to the forum for therapist feedback. The purpose of the therapist responses is to reinforce the development of multiple strategies and help supplement or reshape those that are concrete, based on a predetermined list of strategies developed for each of the computer exercises.
Behavioral: Bridging strategies — The online forum will have illustrations for bridging cognitive abilities and problem solving strategies related to each game to experiences in the real world. An at home workbook will also be used to facilitate active application of skills in various domains (e.g., work, socialization, recreation, household maintenance).

SUMMARY:
Major depressive disorder is the number one cause of disability worldwide. Evidence regarding the effectiveness of various treatments for patients with severe depression is still lacking. Although many patients achieve treatment response, only a minority of patients achieve full remission and even fewer sustain it. In fact, within one month 10% will be re-hospitalized and the rate climbs to 30% within a year. Further, remission from depressive symptoms is a surprisingly poor predictor of recovery of community functioning following discharge. It is clear that the traditional focus on diagnostic symptoms is insufficient for promoting a full return to everyday functioning. The present aim is to examine the efficacy and effectiveness of treating neurocognition, a symptom that explains persistent deficits in community functioning for those with depression. The study design that maps on to the contemporary clinical setting, in order to reflect the changing landscape of inpatient and community treatment.

DETAILED DESCRIPTION:
Cognitive impairment in depression has emerged as one of the most robust predictors of sustained impairment in everyday functioning. Significant deficits in attention, memory and executive function are widespread and remain even after effective treatment of primary mood symptoms. Relevant to the investigators aims, severity of cognitive impairments has been linked to more severe episodes and higher rates of relapse. Cognitive Remediation (CR) is a psychological treatment developed and tested in research settings, where techniques that train the brain to process information more efficiently result in improvements in cognition and in community functioning. Contemporary CR relies on three pillars of treatment: Drill and Practice, Strategic Monitoring, and Bridging of Cognitive Skills to Everyday Life. CR treatment produces robust effects in depression, with some evidence for transfer to reduced depressive symptoms. However, each of the three pillars is typically done within a group therapy context, with two or more meetings per week, presenting a challenge to both modern health care models and the symptoms of depression that would be barriers to attendance (low motivation, social anxiety, lack of energy). The investigators have recently developed a Remote Cognitive Remediation program that overcomes these obstacles with novel components of CR to allow for delivery of treatment remotely. These techniques include the use of online exercises for an increased dose, and the delivery of recorded visual examples of bridging strategies. Efficacy (cognitive improvement) and effectiveness (improved community functioning, reduced time to relapse) will be compared to a placebo control group in this 12-week randomized controlled trial with 6-month follow-up assessments.

This project has the potential to address a significant gap in the treatment of depression and to modify an established treatment to fit into the changing demands of the health care system.

Aim 1: To examine whether cognitive remediation, delivered at home over the Internet, is efficacious in improving cognition in symptomatic individuals with recurrent MDD.

Aim 2: To examine the effectiveness of remote cognitive remediation for improving community functioning.

Aim 3: To examine the baseline and dynamic predictors and mediators of change in functioning for patients with MDD who receive cognitive remediation.

Exploratory Aim: To examine whether cognitive remediation affects rates of response, remission, and relapse.

Hypothesis 1: Remote cognitive remediation will improve neurocognitive functioning at post-treatment and these improvements will persist for 24 weeks.

Hypothesis 2a: Remote cognitive remediation will improve functional capacity at post-treatment and these improvements will persist for 24 weeks.

Hypothesis 2b: Remote cognitive remediation will improve functioning in the community 24 weeks post-treatment.

Hypothesis 3: Improvements in cognitive functioning will predict improvements in functional capacity and functional behaviours post-treatment and 24 weeks later, controlling for depressive symptoms at baseline and change in depressive symptoms. Social cognitive functioning and social anxiety will mediate the degree to which cognitive and functional capacity relate to real world behavior change.

Exploratory Hypotheses:

A.Remote cognitive remediation will increase response and remission rates, and reduce rates of relapse over a 24 week period.

B.12 weeks of CR will demonstrate equivalency in treatment effects to 24 weeks of CR

Participants will be randomized to one of three groups. Two groups will receive active cognitive remediation, with one terminating sessions after 12 weeks (the standard length of time in the literature) and one continuing for a total of 24 weeks of treatment. The third group will receive a comparison training group where they will login to the same training environment but the difficulty level of the working memory load will not progress over time but the tasks will be longer (referred to in the consent as 'focusing your attention for longer periods of time). In previous work, the investigators have found participants to be equally compliant with these groups and for specific changes in memory or attention depending on the group to which they are assigned. Participants will be tested at baseline, 12 weeks (post-intervention, intermediate intervention, or sham, respectively), and at 6 months post-intervention. This design will allow the investigators to test a 2:1 ratio of participants in active memory training versus comparison on the baseline to 12 week assessments and a 1:1:1 comparison for the short-term treatment, long-term treatment, and comparison condition.

Assessments:

Standardized testing will be performed at baseline and/or screening, during clinic visits, and immediately following 12 weeks of intervention. The investigators will also perform a durability assessment at endpoint (end of study participation or at time of dropout) and at 6 months post-treatment to examine the persistence and transfer of effects.

Neurocognition will be assessed with the CNS Vitals system (CNSVS).

Social Cognition will be examined as a potential mediator of changes in cognition and functional capacity to functional behaviour.

The investigators will use the Bell-Lysaker Emotion Recognition Test, which they have previously found to be sensitive to impairment and cognitive treatment in depression.

Functional capacity will be assessed with the Virtual Reality Functional Capacity Assessment, which is a computerized performance based assessment of independent living skills such as planning and shopping.

The 4-item Perceived Competence Scale will assess self-ratings of ability on the measures prior to and after testing.

Functional Behaviour will be assessed with the the World Health Organization Quality of Life Assessment (WHOQoL-BREF).

The Sheehan Disability Scale (SDS) will be used to assess subjective quality of life. The Lam Employment Absence and Productivity Scale (LEAPS) will be used to measure occupational functioning.

Symptoms of depression will be assessed with Montgomery-Asberg Depression Rating Scale MADRS, a gold standard interview-based assessment of 10 items common to MDD.

Other measures that are used include: The Self-Report of Cognitive Lifestyle, The Need for Cognition Scale, The Cognitive Approach Scale, and The Cognitive Failures Questionnaire.

Intervention:

The study will include the foundational Pillars of CR, but modified for this study in a structure that fits contemporary health care systems and with the intention of extending cognitive effects to improved community functioning. The novel components of CR in this study will be the delivery of treatment remotely, the use of online exercises for an increased dose, and the delivery of recorded visual examples of strategic monitoring and bridging strategies.

Pillar I: Cognitive Activation. In the treatment, the use of online exercises allow for a steadier dose of treatment compared to week to week in-person meetings, essential for motivation and learning. There are 30 unique cognitive exercises in the program (sbtpro.com). The investigators will prescribe 24 exercises in the domains most commonly impaired in MDD: six targeting executive functions, ten targeting memory, and eight targeting attention and working memory. The specific activities are prescribed in a fixed, systematic order, such that the participants have a schedule of exercises that address several different cognitive domains each week and return to exercises in subsequent weeks. Parameters are automatically adjusted based on participant performance across 30 difficulty levels. Participants are prescribed two 20-minute sessions per day, five days per week, for the duration of the study. Participants who do not complete tasks for three consecutive days will receive reminder calls from a therapist to address technical or motivational issues.

Pillar II: Strategy Monitoring, Development, and Pruning. Therapists communicate with participants in asynchronous private and group forums, where specific responses to questions prime flexible strategy formation, monitoring of strategies, and bridging to real world functioning. Participants use logs to track their own strategies and upload this information to the forum for therapist feedback. The purpose of the therapist responses is to reinforce the development of multiple strategies and help supplement or reshape those that are concrete, based on a predetermined list of strategies developed for each of the computer exercises.

Pillar III: Bridging. The online forum will have illustrations for bridging cognitive abilities and problem solving strategies related to each game to experiences in the real world. An at home workbook will also be used to facilitate active application of skills in various domains (e.g., work, socialization, recreation, household maintenance).

Comparison Control Group: Comparison cognitive remediation treatment procedures include the same stimuli that are presented in the active treatment condition, but the parameter adjustments change without increasing cognitive demand.

Those who consent will be assigned to the CR or Comparison treatment conditions on a 2:1 basis, based on a computerized random number generator. Allocation to active treatment at 2:1 has advantages related to within group analysis to predict outcomes, trial costs, expected dropouts, and patient acceptability, and does not reduce power. Participants will meet with a study therapist for an orientation to the computer tasks and goal setting in a one-hour training session. Those who experience difficulty understanding or utilizing the program will receive additional training, though this contact will continue to be only computer skill training rather than therapeutic. The study coordinator and assistant will remain available throughout the study for asynchronous responses to email and live telephone support related to usage issues. The goal setting session follows the investigator's standard protocol, which is a collaborative discussion to identify real world functional goals, discuss how the patient's individual cognitive profile links with those goals, and demonstrate how the treatment techniques are related to their profile and everyday functional goals. Ph.D.-level psychology students or psychologists from the PI's laboratory will be available on an asynchronous nature to respond to online Strategic Monitoring and Bridging forum questions and to moderate comments.

ELIGIBILITY:
Inclusion Criteria: Participants must have a primary diagnosis of Major Depressive Disorder

Exclusion Criteria: Medical conditions that affect central nervous system functioning, substance abuse within the past three months (assessed with the SCID-V), and sensory or perceptual conditions that affect validity of testing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-07 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Changes in composite neurocognition scores from the CNS Vitals Signs battery | Participants will be tested at baseline, and assessed for changes at 12 weeks (post-intervention, intermediate intervention, or sham, respectively), and assessed for changes at 6 months post-intervention.
  Neurocognitive Measure

SECONDARY OUTCOMES:
Virtual Reality Functional Capacity Test | Participants will be tested at baseline, and assessed for changes at 12 weeks (post-intervention, intermediate intervention, or sham, respectively), and assessed for changes at 6 months post-intervention.
  Functional Capacity Measure
Composite neurocognition score from the CNS Vitals Signs battery | Participants will be tested at baseline, and assessed for changes at 12 weeks (post-intervention, intermediate intervention, or sham, respectively), and assessed for changes at 6 months post-intervention.
  Functional Capacity Measure
World Health Organization Quality of Life | Participants will be tested at baseline, and assessed for changes at 12 weeks (post-intervention, intermediate intervention, or sham, respectively), and assessed for changes at 6 months post-intervention.
  Everyday Functioning Measure
Bell-Lysaker Emotion Recognition Task | Participants will be tested at baseline, and assessed for changes at 12 weeks (post-intervention, intermediate intervention, or sham, respectively), and assessed for changes at 6 months post-intervention.
  Social Cognition Measure
Montgomery-Asberg Depression Rating Scale | Participants will be tested at baseline, and assessed for changes at 12 weeks (post-intervention, intermediate intervention, or sham, respectively), and assessed for changes at 6 months post-intervention.
  Mood symptom rating
Sheehan Disability Scale | Participants will be tested at baseline, and assessed for changes at 12 weeks (post-intervention, intermediate intervention, or sham, respectively), and assessed for changes at 6 months post-intervention.
  Self-reported quality of life
Lam Employment Absence and Productivity Scale | Participants will be tested at baseline, and assessed for changes at 12 weeks (post-intervention, intermediate intervention, or sham, respectively), and assessed for changes at 6 months post-intervention.
  Work outcomes
Need for Cognition Scale | Participants will be tested at baseline, and assessed for changes at 12 weeks (post-intervention, intermediate intervention, or sham, respectively), and assessed for changes at 6 months post-intervention.
  Self-reported need for cognitive demand in life

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Bowie, Ph D CPsych, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No